CLINICAL TRIAL: NCT01265576
Title: A Randomized, Double Blind, Placebo Controlled, Multicenter Phase 2 Study of VT-122 in Combination With Sorafenib Compared to Sorafenib With Placebo in Patients With Hepatocellular Carcinoma and Systemic Inflammation at Risk for Cachexia
Brief Title: Study of Sorafenib With or Without VT-122 in Patients With Hepatocellular Carcinoma (HCC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VT1-CAX-200
Record Dates: First submitted 2010-12-21; First posted 2010-12-23 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: HCC
MeSH Terms: interventions — Sorafenib; Propranolol; Etodolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib with placebo (Placebo Comparator): Participants randomized to the Control Arm (sorafenib with placebo) receive sorafenib as the standard of care, and placebo for the same periods as participants randomized to the Treatment Arm (sorafenib plus VT-122). Participants randomized to the Control Arm will undergo the same visits and procedures as would the participants randomized to the Treatment Arm.
  Interventions: Drug: Sorafenib; Drug: Placebo
- Sorafenib plus VT-122 (Experimental)
  Interventions: Drug: Sorafenib; Drug: VT-122 (propranolol plus etodolac)

INTERVENTIONS:
Drug: Sorafenib — Participants will be on sorafenib at least 30 days before randomization into either the Treatment or Control Arms. Sorafenib will be administered according to the package insert unless contraindicated based on physician expertise.
Drug: VT-122 (propranolol plus etodolac) — Participants randomized to the VT-122 regimen (sorafenib plus VT-122) will receive oral doses of propranolol and etodolac, which will be titrated over a period of 3 weeks until the participant reaches a maximum tolerated dose (MTD)[no higher than 60 mg propranolol, twice daily (BID)/300 mg etodolac, BID]. Once the individual MTD has been reached, participants will enter a Maintenance Treatment period, and will receive the VT-122 regimen (propranolol and etodolac, co administered orally) on a continuous BID dosing schedule for a maximum of twelve 4-week cycles.
  Arms: Sorafenib plus VT-122
Drug: Placebo — Participants randomized to the Control Arm (sorafenib with placebo) will receive placebo for the same periods as participants randomized to the Treatment Arm. Participants in the Control Arm will undergo the same visits and mock dose escalation.
  Arms: Sorafenib with placebo

SUMMARY:
The purpose of this study is to determine if VT-122 provides a clinical benefit when added to Sorafenib in patients with advanced hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
The most common clinical course of the patient with cancer is local tumor progression leading to the development of metastases, systemic inflammation and the ensuing symptom cluster known as anorexia-cachexia syndrome. This syndrome includes cachexia (anorexia, weight loss and muscle wasting), fatigue, weakness, pain, dyspnea, nausea, malaise, depression and poor performance status. Patients suffering from this syndrome also have poor tolerance, adherence and response to anti-cancer therapy, resulting in disease progression and reduced life expectancy. In spite of the dire need, no proven options for treating inflammatory cancer cachexia are currently available.

VT-122 is the co-administration of the cyclo-oxygenase 2 (COX-2) inhibitor, etodolac and the beta-adrenergic antagonist, propranolol.

It is proposed that these drugs can attenuate systemic inflammation and ameliorate the symptoms of inflammatory cachexia in patients with advanced cancer. As a result, this treatment may improve tolerability and adherence to anti-cancer therapy, thereby yielding direct and indirect benefits in reducing disease progression and improving both the life expectancy and quality of life for patients with advanced cancer.

The potentially synergistic activities of beta blockers and COX-2 inhibitors, their offsetting side effects and their known beneficial impact on co-morbidities associated with liver failure may make them well-suited for use with sorafenib, the standard of care for patients with advanced HCC.

The purpose of this study is to assess whether use of VT-122 is safe and effective in cachectic patients with advanced HCC. In addition to assessing cachexia-related symptoms, the ability of the VT-122 regimen to improve tolerability to sorafenib and thereby to improve both survival and quality of life will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

Participants will be required to meet all of the following criteria to be considered eligible for the study:

* Have a confirmed diagnosis of HCC. Biopsy is preferred but is not required.
* Male and female participants who are ≥18 years of age.
* In the opinion of the investigator, the participants have a life expectancy of at least 12 weeks.
* Able to take food or nutritional support orally.
* On sorafenib for at least 4 weeks prior to randomization. Dose adjustments are allowed prior to randomization.
* Have a Karnofsky Performance Score (KPS) equal to or greater than 50.
* Have a cirrhotic status of Child-Pugh Class A or B7.
* Have the following laboratory parameters:

  * a. Platelet count ≥50 x 10E9/L.
  * b. Total bilirubin ≤1.5 mg/dL (≤1.0 mg/dL for primary biliary cirrhosis). If total bilirubin >1.5 mg/dL but <3.0 mg/dL, a patient could be enrolled after consultation with the Medical Monitor. If total bilirubin is >3.0 mg/dL, but the value has been constant for a period of greater than 3 months, a patient could be enrolled after consultation with the Medical Monitor.
  * c. Serum creatinine ≤1.5 x upper limit of normal (ULN) or creatinine clearance >60 mL/min calculated using Cockcroft-Gault.
  * d. Serum albumin ≤3.5 g/dL and/or C-reactive protein (CRP) ≥3 mg/L
* Able to provide written informed consent prior to any study specific screening procedures with the understanding that the patient has the right to withdraw from the study at any time, for any reason without prejudice.

Exclusion Criteria:

Participants must not have any of the following criteria to be considered eligible for inclusion in the study:

* The patient has a history of another primary cancer, with the exception of: a) curatively resected non-melanomatous skin cancer; b) curatively treated cervical carcinoma in-situ; or c) other primary solid tumor with no known active disease present that in the opinion of the investigator will not affect patient outcome in the setting of current HCC diagnosis.
* Contraindication to sorafenib, propranolol, etodolac, or placebo.
* Patient currently on beta-blockers for the treatment of portal hypertension or arrhythmia. [Patients on beta blockers for the treatment of hypertension are allowed if they change to a different drug class, e.g. some classes of angiotensin-converting enzyme (ACE) inhibitors, for controlling hypertension at least one week before randomization].
* Body mass index (BMI) <17.5 kg/m2.
* History or evidence of cardiac disease: congestive heart failure; New York Heart Association class 2 or greater; active coronary artery disease; unstable angina, cardiac arrhythmias requiring anti-arrhythmic therapy, atrioventricular block of second or third degree, or uncontrolled hypertension. Patients with recent (less than 6 months) myocardial infarction (MI) or coronary revascularization.
* Hypotension at the time of screening (i.e., systolic blood pressure <90 mmHg, diastolic blood pressure <60 mmHg).
* Resting heart rate <60 bpm at time of screening.
* Participants with a recent diagnosis of bleeding varices that has not been resolved for a minimum period of 4 weeks.
* Any uncontrolled intercurrent illness that, in the opinion of the Investigator, may interfere with study evaluation.
* On chronotropic drugs (acetylcholine, digoxin, diltiazem, verapamil, atropine, dopamine, dobutamine, epinephrine, isoproterenol).
* Active clinically serious infections [>Grade 2 National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 4.0].
* Known history of human immunodeficiency virus (HIV) infection.
* Known central nervous system tumors including metastatic brain disease.
* Clinically significant gastrointestinal (GI) bleeding within 30 days prior to Screening.
* Substance abuse, medical, psychological or social conditions that may, in the in the opinion of the investigator, interfere with the patient's participation in the study or evaluation of the study results.
* Known or suspected allergy to the investigational agents or any agent given in association with this trial (hypersensitivity reaction, hives, rash, difficulty breathing swelling of face, lips, tongue, or throat).
* Inability to swallow oral medications.
* Any condition that is unstable or which in the opinion of the Investigator could jeopardize the safety of the patient and his/her compliance in the study.
* Pregnant or breastfeeding participants. Women of childbearing potential (non-childbearing potential is defined as menopausal for at least 2 years, post-bilateral tubal ligation for at least 1 year, post-bilateral oophorectomy or post-hysterectomy) must have a negative urine pregnancy test performed within 10 days prior to the start of study drug. Both men and women enrolled in this trial must use adequate double-barrier birth control measures [2 types of an acceptable form of FDA-approved contraception (e.g., barrier method, Depo-Provera™, Norplant™, Ortho Evra® [birth control patch], oral contraceptives)] during the course of the trial.
* Participation in any other investigational trial in which receipt of investigational drug or device occurred within 30 days prior to screening for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-12; Primary Completion 2014-02 (Actual); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
failure free survival | 6 months

SECONDARY OUTCOMES:
clinical benefit response | 6 months

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Vicus Clinical Site, Berkeley, California
  - Vicus Clinical Site, Atlanta, Georgia
  - Vicus Clinical Site, New Brunswick, New Jersey
  - Vicus Clinical Site, Newark, New Jersey
  - Vicus Clinical Site, Paterson, New Jersey
  - Vicus Clinical Site, Buffalo, New York
  - Vicus Clinical Site, New York, New York
  - Vicus Clinical Site, Philadelphia, Pennsylvania
  - Vicus Clinical Site, Houston, Texas